CLINICAL TRIAL: NCT06496906
Title: Clinical and Radiographic Comparison of Two Minimally Invasive Tooth Extraction Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPDP02/2021
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Tooth Extraction Status Nos
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Benex tooth extraction (Experimental): This is the first study group where patients undergo extractions with presumably the vertical tooth extraction system Benex.
  Interventions: Procedure: Tooth extraction; Device: Benex
- Physics forceps extraction (Experimental): This is the second study group where patients undergo extractions with the presumably minimally invasive Physics forceps.
  Interventions: Procedure: Tooth extraction; Device: Physics Forceps
- Convetional extraction (Active Comparator): This is the control group where patients undergo tooth extractions with conventional extraction forceps and elevators.
  Interventions: Procedure: Tooth extraction; Device: Conventional Extraction Forceps

INTERVENTIONS:
Procedure: Tooth extraction — A regular closed tooth extraction was performed with the different devices from each arm.
Device: Benex — Benex was used to perform the intervention.
  Arms: Benex tooth extraction
Device: Physics Forceps — Physics forceps were used to perform the intervention.
  Arms: Physics forceps extraction
Device: Conventional Extraction Forceps — Conventional Extraction Forceps were used to perform the intervention.
  Arms: Convetional extraction

SUMMARY:
The aim of the study is to compare the effectiveness of the vertical extraction system Benex and Physics forceps with the conventional extraction tools (extraction forceps and elevators) in the early wound healing period after tooth extraction, as means for minimally invasive tooth extraction.

All patients aged 18 years and over who require closed tooth extraction with good oral hygiene were eligible for participation.

Participants were randomly allocated to tooth extraction with either Benex, Physics forceps or conventional extraction tools using box randomization. Patients are followed up during the recovery period to assess pain and early wound healing, while at the time of extraction, success and buccal cortical plate fracture were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with teeth indicated for closed extraction
* Teeth with at least 1mm of tissue above the bone level
* Patients without contraindications for surgical intervention (ASA 1 or 2)
* Patients with good oral hygiene

Exclusion Criteria:

* Patients with severe systemic conditions or immunosuppression
* Teeth with mobility greater than Grade 1
* Teeth indicated for open surgical extraction
* Patients with acute odontogenic infections
* Drug or alcohol abuse
* Patients with psychiatric conditions
* Patients on anticoagulant or antiaggregant drugs refusing to undergo prior tests and preparation for tooth extraction
* Patients on chemotherapy, radiotherapy, or oral bisphosphonate intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Extraction success | From the beginning of the extraction to the completion of the procedure
  The scale suggested by Choi was used to assess each of the extraction systems.
  Scored from 1 to 5. Higher is better.
Alveolar bone buccal cortical plate preservation | From the beginning of the extraction to the completion of the procedure
  The difference between the height of the alveolar bone buccal cortical plate is measured before and after the tooth extraction.
  Scored in milimeters missing. Lower is better.
VAS pain score | 0, 1, 3, 7 day
  Patients were asked to rate their pain experience on a visual analog scale (VAS).
  Measured in centimeters on 10cm line. Lower is better.
Early wound healing | 3, 7, 10 day
  Landry's early wound healing index was used to evaluated the extraction healing process.
  Scores from 1 to 5. Higher is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Surgery, Faculty of Dental Medicine, Medical University - Plovdiv, Plovdiv, Pl, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided